CLINICAL TRIAL: NCT01007214
Title: Hybrid Imaging Technique (HIT) Guided Biopsy to Map Prostatic Adenocarcinoma in Patients Undergoing Prostatectomy
Brief Title: Guided Biopsy for Mapping Prostate Cancer
Acronym: HIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to meet accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 133608
Record Dates: First submitted 2009-10-29; First posted 2009-11-03 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate cancer (Experimental): A total of 30 patients diagnosed with prostate cancer who have elected to undergo radical prostatectomy are enrolled over a six year period.
  Interventions: Procedure: Prostatectomy

INTERVENTIONS:
Procedure: Prostatectomy — Elective prostatectomy
  Other Names: Prostate cancer

SUMMARY:
Evaluate the accuracy of HIT guided biopsies for mapping tumor foci with men undergoing prostatectomy.

DETAILED DESCRIPTION:
The objective of this study is to determine the accuracy of HIT (Hybrid Imaging Technology) guided biopsies for mapping tumor foci with men undergoing prostatectomy. Using a prostate hybrid imaging technology (HIT) which fuses a previously obtained endorectal MR image to transrectal ultrasound (TRUS) image to allow identification and biopsy of tumors by MR imaging in real time. We hypothesis that HIT guided biopsies will accurately localize the foci of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of prostate cancer
* Patients must have elected to undergo radical prostatectomy using an open, laparoscopic or robotic approach
* Patients must be at least 18 years of age and able to provide written informed consent.
* No history of radiotherapy, chemotherapy or hormone therapy within 6 months of surgery
* Primary tumor must be amenable to surgical removal for curative intent
* Patients must have ECOG-performance status 0 or 1 (appendix II)
* Patients must have no history of rectal or anal disease.
* Patients must have adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT])≤2.5x local laboratory upper limit of normal (ULN), or AST and ALT ≤5x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin ≤1.5 x ULN
  * Absolute neutrophil count(ANC)≥1,500/microL
  * Platelets≥lOO,OOO/microL
  * Hemoglobin≥9.0 g/dL
  * Serum calcium≤10.2mg/dL (correct for low albumin if necessary; calcium + (normal albumin - serum albumin)x 0.8)
  * Patients must have serum creatinine<2 mg/dL or serum creatinine clearance (CrCl)>40ml/min(CrCl= Wt(kg)x(140-age)*/72xCr. level,*female x 0.85)

Inclusion of minorities:

* Members of all races and ethnic groups are eligible for this trial. Women and children are not eligible since prostate cancer is not diagnosed in these groups.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Determine the accuracy of hybrid image technology (HIT) guided biopsies for prostate cancer mapping. | Six years

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, MD, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States